CLINICAL TRIAL: NCT06748651
Title: Evaluation of Allocetra by Intra-articular Injection for the Treatment of Temporomandibular Joint Osteoarthritis (TMJ-OA)
Brief Title: Intra-articular Allocetra in Osteoarthritis of the of the Temporomandibular Joint (TMJ)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Amit Druyan (Other Government)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Amit Druyan, Principal Investigator, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1400-24-SMC
Record Dates: First submitted 2024-12-13; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Temporomandibular Joint Osteoarthritis
Keywords: ALLOCETRA; Temporomandibular; Osteoarthritis; TMJ; Macrophages; Cell therapy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: The study will consist of two stages, during which a single treatment of Allocetra, will be administered via intra-articular injection into the target temporomandibular joint .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intra-articular Injection of Allocetra performed once on Day 1 of the study (Experimental)
  Interventions: Drug: Allocetra

INTERVENTIONS:
Drug: Allocetra — Intra-articular injection of Allocetra performed once on Day 1 of the study

SUMMARY:
This study is a single center trial to assess the safety and initial efficacy of intra-articular administration of Allocetra to patients with Temporomandibular Joint Osteoarthritis (TMJ-OA)

DETAILED DESCRIPTION:
The temporomandibular joint (TMJ) is a critical synovial joint enabling jaw movement. TMJ osteoarthritis results from factors such as disc dislocation, trauma, overuse, or developmental anomalies, affecting all joint structures, including cartilage, synovium, bone, and ligaments. Key pathological features include chondrocyte loss, extracellular matrix degradation, and subchondral bone remodeling. TMJ-OA progresses gradually through phases of activity and remission, ultimately leading to a burnout phase.

Allocetra is an immunomodulatory cell-based therapy consisting of allogeneic peripheral blood mononuclear cells that have been modified to be engulfed by macrophages and reprogram them into their homeostatic state.

This study is a single center, open lable safety and initial efficacy trial to assess intra-articular administration of Allocetra in patients with TMJ-OA who have not responded sufficiently to conventional therapies.

The study is comprised of two stages, during which a single treatment of Allocetra, will be administered via intra-articular injection into the target temporomandibular joint.

Patients will be followed for up to a year following treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with temporomandibular OA in the target TMJ.
2. Inflammatory findings by Magnetic Resonance Imaging (MRI).
3. Acceptable blood workup results (CBC, electrolytes, kidney and liver function).

Exclusion Criteria:

1. Prior intra-articular injection to the target TMJ within 3 months prior to treatment.
2. Any significant injury or surgery to the target TMJ.
3. Evidence of active local infection in the vicinity of the target TMJ or clinically significant active infection anywhere in the body.
4. Patients with a known neurological disease or rheumatic condition, a major medical condition that would affect quality of life and influence the results of the study, or other pain of unknown etiology.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2026-02-07 (Estimated); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
Number and severity of AEs, SAEs and injection reactions following treatment | Day 0 to 12 month
  Number and severity of AEs, SAEs and following treatment, and injection-related reactions occurring during study treatment injection, including injection interruption/discontinuation.

SECONDARY OUTCOMES:
Patient reported pain in the target TMJ | Screening to 6 months
  Change from baseline in patient reported pain Numerical Rating Scale (NRS) in the target TMJ at 3 months and 6 months following treatment.

OTHER OUTCOMES:
Exploratory outcome: Assessment of TMJ function by examination | Screening to 12 months
  Number of patients with pain on palpation, clicking/crepitation, or mandibular mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel